CLINICAL TRIAL: NCT06121310
Title: Evaluation of Satisfaction Levels of Pediatric Patients and Parents After Anesthesia: A Turkish Validity and Reliability Study
Brief Title: Turkish Validity and Reliability Study of Pediatric Anesthesia Satisfaction Scale
Acronym: TVRPAS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Yesim Senayli, Assistant Professor, Bozok University
Other Study IDs: Bozok University
Record Dates: First submitted 2023-08-25; First posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pediatric Anesthesia
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Survey grup: No intervention is to be administered. Just a survey study
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Non interventional. Pediatric anesthesia satisfaction scale validity and reliability is going to investigate by survey analyses

SUMMARY:
Strategies to increase patient satisfaction have a positive effect on clinical care. Therefore, evaluation of emotional and psychological satisfaction and satisfaction can increase the quality of anesthetic care. The number of satisfaction evaluation studies, especially for pediatric patients who have undergone surgery, is very few, and the validity and reliability of the existing satisfaction scoring systems in the Turkish population has not yet been established. As a result of this study, it will be possible to use a Turkish validity and reliability scale that can evaluate the satisfaction levels of pediatric patients and parents after anesthesia, which is planned to be developed, to be used in the studies of improving health services, increasing the quality of the hospital, and using it in scientific studies by researchers and academicians in Türkiye.The aim of this study is to conduct a Turkish validity and reliability study by examining the reliability, validity, acceptability and reproducibility of a pediatric patient and parent satisfaction questionnaire previously validated in English.

The research data will be realized by the face-to-face filling of the Turkish version of the pediatric anesthesia satisfaction scale, which has been published in the literature, by the child and their parents.

The Turkish version of the scale in question will be asked to fill out the questionnaire within the first hour of being transferred from the operating room to the pediatric surgery service after the surgery/surgical procedure for all parents who have been operated by Yozgat Bozok University Research and Practice Hospital Pediatric Surgery. The delivery of the questionnaire and its face-to-face filling process will be carried out by an anesthesiologist (specialist or specialist student) different from the relevant anesthesiologist, who is responsible for the outpatient evaluation of the patient and the anesthesia management in the peroperative period, so that the respondent is not affected by any embarrassment, intentional reasons, etc.

ELIGIBILITY:
Inclusion Criteria:

1. Speaking Turkish of the child patient and the parent
2. Absence of any known psychiatric disease
3. Agreeing to participate in the study (patients and parents with cognitive development who can give consent)

Exclusion Criteria:

1. Having any known psychiatric disease of the child patient or parent
2. Having a history of drug use that will affect the cognitive functions of the child patient or parent
3. Parent's refusal to participate in the study (patients and parents with cognitive development who can give consent)
4. Child patient or parent does not know Turkish

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 0-18 years old age pediatric patients who 0-18 year who will undergo surgical procedure
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-15 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Valid and reliable Turkish pediatric anesthesia satisfaction scale | One year
  The reliability, test-retest reliability, and internal consistency will be examined. McNemar coefficient and a Cronbach's alpha coefficient will be applied to get validity conformation

CONTACTS AND LOCATIONS:
Overall Officials: Yesim Senayli, ass profess, Principal Investigator — Bozok University Anesthesiology and Reanimation Department
Locations (1):
- Bozok University, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No